CLINICAL TRIAL: NCT04410822
Title: Fecal Incontinence Type Assessment Scale (FITAS): a New Tool to Distinguish Among Subgroups of Fecal Incontinence
Brief Title: Fecal Incontinence Type Assessment Scale
Status: Completed | Type: Observational
Sponsor: Gérard Amarenco (Other)
Responsible Party: Sponsor-Investigator, Gérard Amarenco, Head of Neuro-Urology Department, Pierre and Marie Curie University
Organization: Pierre and Marie Curie University (Other)
Other Study IDs: GREEN GRC01 FITAS
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Faecal Incontinence
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients enrolled: an age older than 18 years old and symptoms of FI according to Rome IV criteria.
  Interventions: Other: Clinical tests

INTERVENTIONS:
Other: Clinical tests — Semi-qualitative interviews and questionnaire FITAS

SUMMARY:
Urge faecal incontinence (FI) and passive FI are the two subgroups of FI described by the International Continence Society. Urge FI is described as "the inability to defer defecation once the urge is perceived for long enough to reach a toilet" and passive FI as "the involuntary leakage of faeces without forewarning". If several validated questionnaires are available for FI, all of these questionnaires were developed to assess FI severity. In literature, there is only a small number of studies that investigated clinical and paraclinical characteristics of the different phenotype of FI. Moreover, there is an heterogenicity in the definitions used for both urge and passive FI among these studies. Lastly, patients with mixed FI were commonly excluded from these studies. It can be established that there is a lack of validate tools to distinguish patients between subgroups of FI.

The aim of the present study was to develop and to validate a new tool in order to investigate and classify patients among the different subgroups of FI (active, passive and mixed) defined by Rome IV criteria.

A monocentric prospective study was conducted in the Neuro-urology Department of a University Hospital. All consecutive patients presenting in the Department with FI between December 2019 and June 2020 were screened for inclusion in the present study. Criteria of inclusion were an age older than 18 years old and symptoms of FI according to Rome IV criteria. Exclusion criteria were anorectal fistula, active inflammatory bowel disease, anorectal malignant tumor not treated, rectal or hemorrhoidal prolapses and specific inability regarding the questionnaire (i.e. cognitive disorders, inability to read and to understand questions).

Phase 1: review of literature and qualitative interviews: To determine the dimensions of the different subgroups of faecal incontinence, a literature review was performed using Pubmed without date limitation until February 2020. The key words used were "active faecal incontinence", "active fecal incontinence", "passive faecal incontinence", "passive fecal incontinence", "urge faecal incontinence", "urge fecal incontinence", "questionnaire", "scale", "score" and "tool". In parallel to this literature review, semi-structured interviews were performed on 20 patients from December 2019 to February 2020. During this phase, a panel expert of 9 neuro-urologists and gastroenterologists was composed. At the term of all interviews, dimensions that were both the most used by patients and the most discriminative among subgroups of FI were included in the questionnaire. Redaction of questions was then performed by the panel expert.

Phase 2: feasibility study: The feasibility study was conducted from February to April 2020 on 30 patients. Each patient was asked to rate each version of the 2 questions with a four-point Likert scale (A: very good, B: good, C: difficult, D: very difficult) regarding acceptance and comprehension of the questions.

Phase 3: validation study: To investigate the psychometric properties of the questionnaire, a validation study was performed from April to June 2020 on 100 consecutive patients. In order to evaluate the FITAS' test reproducibility, patients were asked to answer a second time the questionnaire by mail with a second evaluation from 7 days to 10 days after the first one. The "intra-class correlation coefficient" (ICC) was used to determine if these evaluations could lead to similar results for each question. An ICC > 0.70 was necessary to define reproducibility.

ELIGIBILITY:
Inclusion Criteria:

* age older than 18 years old
* symptoms of FI according to Rome IV criteria

Exclusion Criteria:

* Anorectal fistula
* Active inflammatory bowel disease
* Anorectal malignant tumor not treated
* Rectal or hemorrhoidal prolapses
* Specific inability regarding the questionnaire (i.e. cognitive disorders, inability to read and to understand questions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting in a tertiary center in neuro-urology
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Reproducibility of FITAS | 1 day
  Patients were asked to answer a second time the questionnaire by mail with a second evaluation from 7 days to 10 days after the first one. The "intra-class correlation coefficient" (ICC) was used to determine if these evaluations could lead to similar results for each question. An ICC > 0.70 was necessary to define reproducibility.
Acceptability of FITAS | 1 day
  Each patient was asked to rate acceptability of FITAS with a four-point Likert scale (A: very good, B: good, C: difficult, D: very difficult) regarding acceptance and comprehension of the questions.
comprehension of FITAS | 1 day
  Each patient was asked to rate comprehension of FITAS with a four-point Likert scale (A: very good, B: good, C: difficult, D: very difficult) regarding acceptance and comprehension of the questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Charlotte Desprez, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided